CLINICAL TRIAL: NCT00136487
Title: A Randomized, Double Blind, Placebo-Controlled Trial of Celecoxib Versus Placebo in Men With Prostate Cancer With Rising PSA Following Prostatectomy or Radiation Therapy
Brief Title: Celecoxib (Celebrex) Versus Placebo in Men With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry); Beth Israel Deaconess Medical Center (Other); Emerson Hospital, Concord, MA (Other); Brigham and Women's Hospital (Other); Hartford Hospital (Other); Lowell General Hospital (Other); Massachusetts General Hospital (Other); M.D. Anderson Cancer Center (Other); University of Michigan Rogel Cancer Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02-193; COXAON-0509-125
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Cancer of Prostate; Cancer of the Prostate; Prostate-Specific Antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
The purpose of this study is to learn the effects (both good and bad) that celecoxib has on prostate cancer and patients with prostate cancer. This study is looking at what effects celecoxib has on prostate specific antigen (PSA) level. PSA is a marker specific to prostate cancer. An increase or decrease in this level in the blood can indicate if a patient's prostate cancer is getting worse or better.

DETAILED DESCRIPTION:
This study is designed as a randomized, double blind, placebo-controlled study. These are all scientific research methods used to protect the study from personal bias or prejudice.

Patients who participate in this study will be randomly assigned initially to take either celecoxib (the study drug) or placebo (an inactive substance that looks like the study drug). Placebos are used to help determine if the results of a study (good or bad) result from chance or from treatment with the study drug. Patients will have a fifty-fifty chance of initial treatment with the study drug. Neither the patient nor the patient's doctor will know whether he/she is initially receiving the study drug or placebo. Participants who are assigned to initially take placebo may have the opportunity to be treated with celecoxib later in the study.

If patients are found to be eligible for this study and they agree to participate, they will be randomized to either receive celecoxib or placebo to be taken by mouth (as a pill) twice a day, every day for as long as they are in the study. Patients will be given a pill diary to keep track of their medications. While in this study, they will be asked not to take any non-steroidal anti-inflammatory drugs, which includes over-the-counter ibuprofen and many other available drugs. In addition, they will be asked not to take any other selective COX-2 inhibitors (the class of drug that celecoxib is).

While in this study, patients will have evaluations (physical exam and blood) to determine their response to their assigned regimen and to monitor side effects.

Once a month the following will be performed:

* Review of any side effects
* Physical Exam
* Routine blood tests (PSA level, kidney function). About one tablespoon of blood will be taken at each visit.

Every other month starting with month 2:

In addition to the above evaluations, on alternating months starting with month 2, additional routine blood tests (liver function, complete blood count) will be done. This will require an additional tablespoon of blood to be taken at these visits.

Additional blood for research-related testing (about 2-3 tablespoons) will also be drawn during these visits.

Participation in this study will be determined by how well patients tolerate the assigned regimen and by how their disease responds. Patients will continue taking their assigned regimen for 6 months as long as it is felt that their disease is stable (based on their PSA levels) and they are tolerating the treatment. After 6 months or earlier, if the disease progresses, the treatment code will be broken. If patients were on celecoxib, they will be taken off study. The patient's doctor will discuss other available treatment options with him/her at that time, including continuing celecoxib "off study". If patients were on placebo, they will then have the option to begin taking celecoxib. If patients start celecoxib treatment, they will be treated in this study with celecoxib for 6 months or until their disease progresses. After 6 months on celecoxib or sooner, if their disease progresses, they will be taken off study. The patient's doctor will discuss available treatment options with him/her at that time, including continuing celecoxib "off study".

Patients who are taken "off study" will be monitored monthly for patient safety reasons throughout the duration of time that they are receiving celecoxib at the dose level used for this study (400mg twice a day).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer
* Progression following prostatectomy or radiation to the prostate, defined as 3 PSA rises, with each PSA determination at least 4 weeks apart
* PSA greater than or equal to 1.0 for men who had a prostatectomy
* PSA greater than or equal to 3.0 for men who were treated with primary radiation therapy (external beam and/or brachytherapy)
* PSA doubling time between 6 and 24 months
* Participants must be either fully active and asymptomatic or symptomatic but fully ambulatory
* Adequate bone marrow function, kidney function and liver function as evidenced by laboratory results

Exclusion Criteria:

* Evidence of metastatic disease
* Prior hormonal therapy for recurrent prostate cancer
* Prior chemotherapy for recurrent or metastatic prostate cancer
* Radiation therapy within 6 months
* Patients allergic to non-steroidal anti-inflammatory drugs (NSAIDs), salicylates or sulfonamide-type medications who experience asthma or urticaria (hives) after taking aspirin or other NSAIDs
* Patients taking a dose of aspirin greater than or equal to 325 mg a day within 4 weeks of study entry
* Patients taking selective COX-2 inhibitors or any NSAIDs other than aspirin within 8 weeks of study entry
* Patients taking fluconazole, lithium or warfarin
* History of gastrointestinal or abdominal ulceration or any history of significant gastrointestinal bleeding in the past 12 months
* Any history of myocardial infarction in the past 12 months
* Any uncontrolled, serious medical or psychiatric illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Start 2002-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the biologic activity of celecoxib by comparing the proportion of men with a post-treatment PSA doubling time (PSADT) greater than or equal to 200% pre-treatment PSADT in the celecoxib-treated group compared to the placebo-treated group

SECONDARY OUTCOMES:
To compare changes in PSADT between the first and second six-month treatment periods for those in the placebo-treated group
to correlate COX-2 expression in the patients' original prostate samples with biologic activity of celecoxib (when feasible)
to correlate changes in plasma vascular endothelial growth factor (VEGF) levels in patients with biologic activity of celecoxib

CONTACTS AND LOCATIONS:
Overall Officials: Philip W. Kantoff, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - Hartford Hospital, Hartford, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Emerson Hospital, Concord, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas